CLINICAL TRIAL: NCT03357965
Title: Evaulation of Maternal-infant Bonding in Postpartum Period of Healthy Women With Family Medicine Perspective
Brief Title: Familiy Medicine Perspective to Maternal-infant Bonding
Status: Completed | Type: Observational
Sponsor: Yildiz Atadag (Other Government)
Responsible Party: Sponsor-Investigator, Yildiz Atadag, Medical Doctor, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Other Study IDs: 18517
Record Dates: First submitted 2017-11-20; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Maternal-Fetal Relations; Depression; Anxiety
Keywords: maternal infant bonding; depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Women who had gave birth in 6 weeks

SUMMARY:
Maternal bonding was described as a qualitative change in the relationship of a mother with her infant. By this study, the investigators aimed to investigate the mother-infant bonding and the factors affecting it, from the point of the family practice, which is responsible for the healthcare of all family members from the fetus to the eldest individual in a family.

DETAILED DESCRIPTION:
The study was carried out as a single-centered descriptive research among 73 women at the postpartum period. The sociodemographic status and the histories of pregnancies of the study participants were recorded. The Maternal Attachment Inventory (MAI), which questions the biological, psychological and social factors, and the Hospital Anxiety and Depression Scale (HADS) were used to collect data to determine the factors affecting the mother-infant bonding in the postpartum period.

The study is a descriptive survey study, which was conducted to determine the mother-infant attachment and its affecting factors in mothers in the first 6-week of the postpartum period. In order to conduct the study, the local Ethics Committee approval was obtained. (Approval date: 24.11.2016, number 18517).

The mean score of the Turkish version of the Maternal Attachment Inventory (MAI) is approximately 95+6 according to the validation study. In our study, considering that the average MAI score of the participants would be approximately 97, investigators determined to include 73 patients in the study with a type I error set at a=0.05 and with the power of (1-b) 80%.

The universe of the study consists of the mothers in the first 6 weeks of the postpartum period presenting to the Obstetrics and Gynecology Clinic and the mothers of the pediatric patients presenting to the Pediatric Clinic of the Health Sciences University Umraniye Education and Research Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Women who gave birth in 6 weeks
* Women who had no mental illness history
* Women who had no health issue
* Women who accepted to join the study
* Women who can communicate

Exclusion Criteria:

* The women who did not have the features below the inclusion criteria

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The universe of the study consists of the mothers in the first 6 weeks of the postpartum period presenting to the Obstetrics and Gynecology Clinic and the mothers of the pediatric patients presenting to the Pediatric Clinic of the Health Sciences University Umraniye Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Maternal Attachment Inventory | 20 minutes
  The items of the MAI are designed in the 4-point Likert scale, which can be scored between 1 and 4 (1: never, 2: sometimes, 3: often, 4: always). The increasing scores indicate increasing levels of attachment of the mother.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Sahinbey Baglarbasi Family Health Center, Gaziantep, Turkey (Türkiye)

REFERENCES:
- [Background] Bowlby J. Attachment and Loss Volume I: Attachment. 2nd ed. New York: Basic Books Inc; 1982
- [Background] Cranley MS. Development of a tool for the measurement of maternal attachment during pregnancy. Nurs Res. 1981 Sep-Oct;30(5):281-4. PMID 6912989
- [Background] BOWLBY J. The nature of the child's tie to his mother. Int J Psychoanal. 1958 Sep-Oct;39(5):350-73. No abstract available. PMID 13610508
- [Background] Bowlby J. Attachment and Loss Volume II: Separation. Anxiety and Anger. New York: Basics Books, Inc; 1973.
- [Background] Rodriguez CM, Tucker MC. Behind the cycle of violence, beyond abuse history: a brief report on the association of parental attachment to physical child abuse potential. Violence Vict. 2011;26(2):246-56. doi: 10.1891/0886-6708.26.2.246. PMID 21780538
- [Background] Kapci EG, Kucuker S. [The parental bonding instrument: evaluation of psychometric properties with Turkish university students]. Turk Psikiyatri Derg. 2006 Winter;17(4):286-95. Turkish. PMID 17183445
- [Background] Noriuchi M, Kikuchi Y, Senoo A. The functional neuroanatomy of maternal love: mother's response to infant's attachment behaviors. Biol Psychiatry. 2008 Feb 15;63(4):415-23. doi: 10.1016/j.biopsych.2007.05.018. Epub 2007 Aug 7. PMID 17686467
- [Background] Pirdal H, Yalçın BM, Ünal M. Knowledge levels of pregnants on their pregnancy and the related factors. Turkish Journal of Family Practice. 2016;20(1):7-15.
- [Background] Atadağ Y, Aydın A, Kaya D, Köşker HD, Başak, F, Uçak S. Changes in causes of admission to tertiary health care center with family medicine implementation. Turkish Journal of Family Practice. 2016;20(4):141-151
- [Background] Aydemir Ö, Güvenir T, Küey L ve ark (1997) Validity and Reliability of Turkish Version of Hospital Anxiety and Depression Scale. Turkish Journal of Pscyhiatry. 8(4): 280-287.